CLINICAL TRIAL: NCT01287208
Title: Be Fit in Residency: a Randomized Controlled Trial of an Activity Device Among Medicine Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anne N. Thorndike, MD, MPH, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-P-001271; 1K23HL093221 (NIH)
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Physical Activity
Keywords: Physical activity; Accelerometer; Steps; Medical residents
MeSH Terms: conditions — Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unblinded activity monitor (Active Comparator): Subjects wear the activity device and can see the data on the device and on a website where the data is uploaded.
  Interventions: Device: Activity monitor
- Blinded activity monitor (Placebo Comparator): Subjects wear a blinded activity device and cannot see the activity on the device and cannot log on to the website where the data gets uploaded.
  Interventions: Device: Activity device

INTERVENTIONS:
Device: Activity monitor — The activity monitor is an accelerometer that records steps, distance, calories, and sleep
  Other Names: Fitbit
  Arms: Unblinded activity monitor
Device: Activity device — Accelerometer that has all the steps, distance, calories, and sleep data blinded to the study subject
  Other Names: Fitbit
  Arms: Blinded activity monitor

SUMMARY:
The main objective of this study is to test an intervention to increase the physical activity of medical residents, an employee population with little time for exercise. Specifically, the aims of this study are:

1. To determine if providing medical residents with an activity device that measures steps, distance, and calories burned and tracks this information over time on a website increases residents' physical activity levels as measured by number of steps per day compared to a control group using a blinded activity device (no feedback).
2. To determine if an unblinded team competition using the activity device directly following the randomized phase increases residents' activity level compared to baseline.
3. To determine if activity level is associated with change in weight during the residency year.
4. To determine if the average hours of sleep per week is associated with changes in weight and with activity level.

ELIGIBILITY:
Inclusion Criteria:

* Massachusetts General Hospital medicine resident

Exclusion Criteria:

* none

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne N Thorndike, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Thorndike AN, Mills S, Sonnenberg L, Palakshappa D, Gao T, Pau CT, Regan S. Activity monitor intervention to promote physical activity of physicians-in-training: randomized controlled trial. PLoS One. 2014 Jun 20;9(6):e100251. doi: 10.1371/journal.pone.0100251. eCollection 2014. PMID 24950218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical residents were recruited during ambulatory care blocks from July 2010 through November 2010.
Pre-assignment Details: Subjects were randomized at the end of December 2010. Four residents withdrew prior to randomization (1 changed mind, 2 said they did not have time, 1 did not complete baseline assessment).
Groups:
- Unblinded: Subjects wear the activity device and can see the data on the device and on a website where the data is uploaded.
- Blinded: Subjects wear a blinded activity device and cannot see the activity on the device and cannot log on to the website where the data gets uploaded.
Period: Phase 1: Randomized Phase
Arm/Group | Unblinded | Blinded
Started | 52 | 52
Completed | 50 | 49
Not Completed | 2 | 3
Period: Phase 2: Team Competition
Arm/Group | Unblinded | Blinded
Started | 50 | 49
Completed | 50 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Unblinded: Activity monitor with visible and on-line feedback
- Blinded: Activity monitor with no feedback
- Total: Total of all reporting groups
Arm/Group | Unblinded | Blinded | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 52 | 104
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (0.3) | 29 (0.4) | 29 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 25 | 23 | 48
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Steps Per Day
Description: Steps will be recorded on the activity device
Time Frame: 12 weeks
Population: We excluded 4 participants who withdrew prior to randomization and 5 who withdrew after randomization.
Measure: Median (Inter-Quartile Range); unit: steps per day
Arm/Group | Unblinded | Blinded
Number analyzed (Participants) | 50 | 49
steps per day | 6369 [1999 to 8796] | 6063 [1299 to 8723]
Statistical Analysis 1: Comparison: Blinded; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Distance Per Day
Description: Distance in miles recorded on activity device.
Time Frame: 12 weeks
Population: This outcome was not collected because of logistical issues with obtaining this data without using an API.
Arm/Group | Unblinded | Blinded
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Calories Burned Per Day
Description: Total calories burned per day recorded on activity device. This secondary outcome was not measured in the trial.
Time Frame: 12 weeks
Population: This outcome was not collected because of logistical issues with obtaining this data without using an API.
Groups:
- Unblinded: Subjects wear the activity device and can see the data on the device and on a website where the data is uploaded.
  Activity monitor: The activity monitor is an accelerometer that records steps, distance, calories, and sleep
- Blinded: Subjects wear a blinded activity device and cannot see the activity on the device and cannot log on to the website where the data gets uploaded.
  Activity device: Accelerometer that has all the steps, distance, calories, and sleep data blinded to the study subject
Arm/Group | Unblinded | Blinded
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Weight
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Unblinded | Blinded
Number analyzed (Participants) | 50 | 49
Pounds | 155 (28.5) | 155 (26.3)
Statistical Analysis 1: Comparison: Unblinded vs Blinded; Test type: Superiority; p = 0.59, t-test, 2 sided

5. Secondary Outcome: Hours of Sleep Per Night
Description: Number of hours slept per night as recorded on activity device.
  This secondary outcome was not measured in the trial.
Time Frame: 12 weeks
Population: This outcome was not collected because of logistical issues with obtaining this data without using an API.
Arm/Group | Unblinded | Blinded
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Unblinded | Blinded
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

LIMITATIONS AND CAVEATS:
Wearing the device may have increased steps in both groups and decreased ability to see a difference.

Unable to collect some secondary outcomes due to logistical issues with obtaining this data without an applications program interface (API).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes